CLINICAL TRIAL: NCT00000175
Title: The Effects of Sex Hormones on Cognition and Mood in Older Adults
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IA0016
Record Dates: First submitted 1999-10-29; First posted 1999-11-01 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2004-03

CONDITIONS: Cognition Disorders; Mood Disorders
Keywords: Emotions; Cognition; Aging; Memory
MeSH Terms: conditions — Cognition Disorders; Mood Disorders | interventions — Estrogens; Testosterone

INTERVENTIONS:
Drug: Estrogen
Drug: Testosterone

SUMMARY:
This study is investigating the effects of hormone replacement therapy on memory, mental abilities and mood in older adults aged 65-90. During the nine month long study, men will take testosterone for three months and women will take estrogen for three months. At four points during the study (once every three months), participants will complete a test battery and have blood drawn.

DETAILED DESCRIPTION:
Double-blind, placebo-controlled, crossover study investigating the effects of estrogen replacement and testosterone replacement on cognition and mood in older adults. Women who have not had a hysterectomy will be given Prempro (estrogen with progesterone to protect the uterine lining), and hysterectomized women will be given Premarin (estrogen only).

ELIGIBILITY:
Inclusion Criteria:

* Women and men aged 65-90 who have not received hormone replacement for the last three months.

Exclusion Criteria:

* Previous head injury with loss of consciousness for more than one hour.
* Men with a history of prostate cancer.
* Men on testosterone replacement within the past three months.
* Women with a history of breast or uterine cancer.
* Women on estrogen replacement within the past three months.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Dates: Primary Completion 2005-06 (Estimated); Study Completion 2005-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Pauline Maki, Principal Investigator — National Institute on Aging, Gerontology Research Center
Locations (1):
- Gerontology Research Center, Baltimore, Maryland, United States

REFERENCES:
- [Background] Henderson VW. The epidemiology of estrogen replacement therapy and Alzheimer's disease. Neurology. 1997 May;48(5 Suppl 7):S27-35. doi: 10.1212/wnl.48.5_suppl_7.27s. PMID 9153164
- [Background] Janowsky JS, Oviatt SK, Orwoll ES. Testosterone influences spatial cognition in older men. Behav Neurosci. 1994 Apr;108(2):325-32. doi: 10.1037//0735-7044.108.2.325. PMID 8037876
- [Background] Sherwin BB. Estrogen effects on cognition in menopausal women. Neurology. 1997 May;48(5 Suppl 7):S21-6. doi: 10.1212/wnl.48.5_suppl_7.21s. PMID 9153163